CLINICAL TRIAL: NCT03048864
Title: Use of Metabolic Evaluations for Patients With Renal Calculi and the Risk of Recurrence
Brief Title: Questionnaire for Metabolic Screening
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Université de Montréal (Other); McGill University (Other); Dalhousie University (Other); University of Toronto (Other); University of Alberta (Other)
Responsible Party: Principal Investigator, Ben Chew, MD, Associate Professor, University of British Columbia
Other Study IDs: H16-03324
Record Dates: First submitted 2017-02-01; First posted 2017-02-09 (Estimated); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Metabolic Evaluation
Keywords: Metabolic Screening; 24 hour urine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to determine if kidney stone patients who should have received metabolic tests (urine collection over 24-hours that determines the composition of urine) based on Canadian Urologic Association (CUA) guidelines did in fact receive them, and if these results were explained to them by their doctor.

DETAILED DESCRIPTION:
PURPOSE:

The purpose of the project is to determine whether metabolic workups are administered to Canadian kidney stone patients in accordance to CUA (Canadian Urologic Association) guidelines. Additionally, the study will look to evaluate whether the results of metabolic tests were sufficiently explained to patients by their doctors, and also whether or not patients would follow dietary or treatment plans to possibly prevent kidney stones based on these metabolic workups.

HYPOTHESIS:

The investigators hypothesize that the implementation of metabolic tests based on CUA guidelines is sub-optimal and that when they are prescribed, doctors do not adequately explain these results to patients. The investigators also hypothesize that patients would follow dietary and treatment plants to prevent recurrent stone formation based on these metabolic results - if they are prescribed to the patient.

JUSTIFICATION:

The investigators believe that implementation of metabolic workups is sub-optimal. The investigators would like to confirm this so that, in the future, metabolic workups can be promoted as an appropriate tool for identifying metabolic abnormalities that contribute to stone disease. If metabolic workups are administered and explained adequately to patients then further diet or treatment plans can significantly reduce recurrence of stones in stone patients.

OBJECTIVES:

1. Determine if metabolic workups were administered when they should have been according to CUA guidelines.
2. For patients who received metabolic workups, determine if the results from metabolic workups were explained to patients, and if so was it done adequately (did the patient understand the explanation)
3. Determine patient compliance regarding dietary and treatment plans based on metabolic workups

RESEARCH DESIGN:

This is a survey based study (one time completion) given to patients pre-ESWL. The surveys will be analyzed by research staff to determine the study objectives.

ELIGIBILITY:
Inclusion Criteria:

* at least 19 years of age, with at least 1 stone episode, ability to consent

Exclusion Criteria:

* inability to provide informed consent, under 19 years of age

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be screened prior to extracorporeal shockwave lithotripsy and will have had at least 1 stone episode. Participants will be recruited from Saint-Luc Hospital, VGH Hospital, Glen Hospital, Dartmouth General Hospital, St.Michael's Hospital and University of Alberta Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-10-27 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Metabolic Evaluation | through study completion - an average of 10 months
  Number of participants that did not receive metabolic evaluations based on Canadian Urologic Association (CUA) criteria

SECONDARY OUTCOMES:
Doctor Patient Communication | at the end of study completion - an average of 10 months
  Number of Participants that received metabolic evaluations but did not have the results adequately explained to them
Patient Dietary/Treatment Compliance | at the end of study completion - an average of 10 months
  Number of patients willing to comply with dietary/treatment advice based on the results of the metabolic evaluations

CONTACTS AND LOCATIONS:
Overall Officials: Nhaeem Bhojani, MD, Principal Investigator — Université de Montréal; Ben H Chew, MD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No